CLINICAL TRIAL: NCT03418350
Title: The Role of Laryngopharyngeal Reflux in IPF
Status: Recruiting | Type: Observational
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Jeff Swigris, Associate Professor, National Jewish Health
Other Study IDs: HS-3130
Record Dates: First submitted 2018-01-23; First posted 2018-02-01 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: IPF; Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to show that the Supraglottic Index (SGI) is an easily-collected index that accurately identifies the presence and severity of laryngopharyngeal reflux (LPF) in idiopathic pulmonary fibrosis (IPF).

DETAILED DESCRIPTION:
The study team hypothesizes the SGI will correlate more strongly with measures of IPF severity (at baseline and over time) than gastroesophageal reflux (GER) data derived from the esophageal detector channels of a pH/impedance probe.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IPF
* Age 40-95
* Able to read, speak, and understand English
* If subjects are currently taking medication for reflux or GERD, they much be on a stable does for at least 4 weeks prior to consent.

Exclusion Criteria:

* Patients who do not meet all inclusion criteria
* Pregnant females

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ILD clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The supraglottic index (SGI) quantifies laryngopharyngeal reflux (LPF) and is associated with severity of pulmonary fibrosis. | 6 months
  Correlation between the supraglottic index and forced vital capacity. The supraglottic index is an index derived by assigning scores for edema and erythema of five supraglottic structures (epiglottis, false cords, arytenoids, posterior commissure, piriform recess) as viewed through a fiber-optic scope. Scores range from 0-22, with higher scores indicating more severe LPR.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Koslow, DO, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be available to other researchers.